CLINICAL TRIAL: NCT05051215
Title: Alterations in the Gut Microbiota and Metabolite Profiles of Nonpuerperal Mastitis Patients
Brief Title: Gut Microbiota and Nonpuerperal Mastitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: Jing Feng 2021-08-15
Record Dates: First submitted 2021-09-06; First posted 2021-09-21 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Microbiota
Keywords: Gut Microbiota; Nonpuerperal mastitis; Plasma cell mastitis; Granulomatous mastitis; Metabonomics
MeSH Terms: conditions — Granulomatous Mastitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — microbiota DNA are extracted from human feces
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: 40 healthy volunteers were included in the healthy control group
- NPM group: 60 patients of NPM (30 PCM and 30 GM)were included

INTERVENTIONS:
Other:

SUMMARY:
Nonpuerperal mastitis (NPM), mainly including Plasma cell mastitis (PCM) and Granulomatous mastitis (GM), which clinical presentation is an accessible and painful breast mass accompanied by skin redness and swelling, nipple retraction and fistula formation . Much progress has been made in exploring the etiology and pathogenesis of NPM, while the exact etiology remains unknown, NPM is thought to arise from interactions between genetic susceptibility factors, epigenetic effects, and various environmental factors. While microbiota as an environment factor to some inflammatory and autoimmune diseases accept widespread attention, if gut microbiota also as a risk factor for NPM, it is worthy to be considered.

DETAILED DESCRIPTION:
NPM is common in young women of reproductive age with a history of lactation and childbearing . The main clinical presentation is an accessible and painful breast mass accompanied by skin redness and swelling, nipple retraction and fistula formation

. The imaging of NPM is not specific, with NPM mimicking breast cancer in imaging . NPM etiology is associated with several factors, such as autoimmunity, bacterial infections , estrogen and progesterone imbalance , and hyperprolactinemia . In recent years, NPM has become a common benign breast disease, especially in the Mediterranean region and developing countries in Asia, such as China . Currently, the associations between bacterial infections and NPM are among the important issues attracting research interest. This study tried to reveal the roles of gut microbiota in NPM. Further understanding of the roles of gut microbiota in this disease may lead to the development of methods for personalized therapy.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 65 years
* Patients of NPM

Exclusion Criteria:

* Pregnancy
* Lactation
* Cigarette smoking
* Alcohol addiction
* Hypertension
* Diabetes mellitus
* Lipid dysregulation
* BMI > 27 <18.5
* Recent (< 1 months prior) use of antibiotics, probiotics, prebiotics, synbiotic, hormonal medication, laxatives, proton pump inhibitors, insulin sensitizers or Chinese herbal medicine
* History of disease with an autoimmune component, such as multiple sclerosis(MS), rheumatoid arthritis, irritable bowel disease(IBS), or irritable bowel syndrome(IBD)
* History of malignancy or any gastrointestinal tract surgery

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study Population are aged from 18 to 65 years#which divided into 2 groups: NPM group and Control group
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-08-15 (Actual); Primary Completion 2023-08-15 (Estimated); Study Completion 2024-08-15 (Estimated)

PRIMARY OUTCOMES:
Microbial profiling of Nonpuerperal Mastitis patients and Healthy controls | Baseline
  16S ribosomal ribonucleic acid(rRNA) gene sequencing technique and illumina MiSeq platform were applied to investigate the difference of gut microbiota richness, diversity and composition between NPM and Healthy controls，and revealing the special gut microbiota profiling data of NPM.

SECONDARY OUTCOMES:
Metabolic profiling of Nonpuerperal Mastitis patients and Healthy controls | Baseline
  Fecal samples were prepared for Ultra-performance liquid chromatography quadrupole time of-flight tandem mass spectrometry (UPLC-Q-TOF/MS) to investigate the difference metabolites and metabolic pathway between NPM and Healthy controls

OTHER OUTCOMES:
Serum Levels of Immune factor | Baseline
  Elisa technique was applied to detect the levels of serum Immune factor (IL-2/IL-4/IL-6/IL-17/IL-10/Lipopolysaccharide) in NPM patients and Healthy controls

CONTACTS AND LOCATIONS:
Overall Officials: Jing Feng, Study Director — First Affiliated Hospital of Harbin Medical University
Locations (1):
- First affiliated hospital of Harbin medical university, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: No